CLINICAL TRIAL: NCT03337074
Title: Investigation of the Effect of Raised Serum Bile Acids on the Epigenome of Sperm and the Association With the Metabolic Health of the Children of Men With Cholestasis: a Case-control Study.
Brief Title: Paternally Inherited Phenotypes in Cholestasis
Acronym: PIP-C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 182833
Record Dates: First submitted 2017-11-01; First posted 2017-11-08 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Cholestasis; Primary Sclerosing Cholangitis; Primary Biliary Cirrhosis
MeSH Terms: conditions — Cholestasis; Cholangitis, Sclerosing; Liver Cirrhosis, Biliary | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sperm Epigenome arm:
  A semen sample and blood sample will be retained for study purposes.
  Outcomes arm:
  A blood sample will be retained for study purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Sperm Epigenome arm/healthy men: Men with no significant health problems.
  Interventions: Other: Questionnaire, semen sample, fasting blood sample
- Sperm Epigenome arm/cholestatic men: Men with a cholestatic liver condition including but not restricted to Primary Sclerosing Cholangitis and Primary Biliary Cholangitis.
  Interventions: Other: Questionnaire, semen sample, fasting blood sample
- Outcomes arm/Cholestatic fathers: Fathers who were diagnosed with a cholestatic liver condition including but not restricted to Primary Sclerosing Cholangitis and Primary Biliary Cholangitis either before or after the conception of their child who is now aged 16 - 25 years of age.
  Interventions: Other: Questionnaire
- Outcomes arm/Children of cholestatic fathers: 16 - 25 years-old children of fathers who were diagnosed with a cholestatic liver condition including but not restricted to Primary Sclerosing Cholangitis and Primary Biliary Cholangitis either before or after their conception.
  Interventions: Other: Questionnaire, fasting blood sample

INTERVENTIONS:
Other: Questionnaire, semen sample, fasting blood sample — Participants are asked to complete a questionnaire and provide a semen sample and fasting blood sample.
  Groups: Sperm Epigenome arm/cholestatic men; Sperm Epigenome arm/healthy men
Other: Questionnaire — Participants are asked to complete a questionnaire.
  Groups: Outcomes arm/Cholestatic fathers
Other: Questionnaire, fasting blood sample — Participants are asked to complete a questionnaire and provide a fasting blood sample.
  Groups: Outcomes arm/Children of cholestatic fathers

SUMMARY:
For some years investigators have known that the health of fathers at the time their baby is conceived has an influence on the health of their child in the future. Many studies looking at this effect have investigated fathers with obesity and other metabolic disorders. These disorders can alter the risk of obesity and diabetes in the children of these men. More recently, studies have been undertaken to establish the mechanism by which this risk is inherited by the children. Studies of sperm have identified that changes in the structure and function of the sperm play a role.

Primary Sclerosing Cholangitis (PSC) and Primary Biliary Cholangitis (PBC) are included in a group of cholestatic liver disorders that are associated with elevated levels of bile acids in the blood (cholestasis). A previous study has established that children born to women who have cholestasis during pregnancy are at an increased risk of obesity later in life. Our study will investigate whether there is a similar effect on the health of children if their father has cholestasis.

The study has 2 arms, the Sperm Epigenome arm and the Outcomes arm.

In the Sperm Epigenome arm of the study, the structure and function of sperm from men with PSC, PBC and other cholestatic liver disorders will be investigated and compared to the structure and function of sperm from healthy men.

In the Outcomes arm of the study, basic health parameters of fathers who had PSC, PBC or another cholestatic liver disease either before or after their child was conceived will be studied. Basic health parameters will also be studied in their child when the child is between 16 and 25 years of age.

ELIGIBILITY:
Sperm Epigenome Arm:

Cholestatic men

Inclusion Criteria:

* Men who have a diagnosis of a cholestatic liver condition including but not restricted to Primary Sclerosing Cholangitis and Primary Biliary Cholangitis.
* Me who are able and willing to give informed consent.

Exclusion Criteria:

* Men who have a history of diabetes or obesity.
* Men who have gallstones, cancer or other acute cholestatic pathology.
* Men who have a history of alcohol excess or drug abuse.
* Men who smoke.
* Men who have blood-borne viruses e.g. HIV or hepatitis.
* Men unable or unwilling to give informed consent

Healthy men

Inclusion Criteria:

* Men who have no history of cholestasis, liver disease, diabetes or obesity.
* Me who are able and willing to give informed consent.

Exclusion Criteria:

* Men who have a history of cholestasis or liver disease.
* Men who have a history of diabetes or obesity.
* Men who have a history of alcohol excess or drug abuse.
* Men who smoke.
* Men who have blood-borne viruses e.g. HIV or hepatitis.
* Men undergoing fertility treatment due to male factor.
* Men unable or unwilling to give informed consent

Outcomes Arm:

Fathers

Inclusion Criteria:

* Fathers with a cholestatic liver condition including but not restricted to Primary Sclerosing Cholangitis and Primary Biliary Cholangitis.
* Fathers with cholestatic liver condition whose children are between 16 years - 25 years of age.
* Fathers with cholestatic liver condition who are able and willing to give informed consent.

Exclusion Criteria:

* Fathers with a history of diabetes or obesity at the time of conception of their child.
* Fathers with a history of alcohol excess or drug-abuse at the time of conception of their child.
* Fathers who smoked at the time of conception of their child.
* Fathers with blood-borne viruses e.g. HIV and hepatitis at the time of conception of their child.
* Fathers unable or unwilling to give informed consent.

Children of cholestatic fathers

Inclusion Criteria:

* Adolescents / young adults (between 16 - 25 years of age) whose fathers have a cholestatic liver condition including but not restricted to Primary Sclerosing Cholangitis or Primary Biliary Cholangitis.
* Adolescents /young adults born from an uncomplicated singleton pregnancy.
* Adolescents /young adults who are able and willing to give informed consent.

Exclusion Criteria:

* Adolescents / young adults who were born as a result of multi-fetal pregnancy.
* Adolescents / young adults with a history of alcohol excess or drug-abuse.
* Adolescents / young adults who are under 16 years of age, or over 25 years of age.
* Adolescents / young adults with blood-borne viruses e.g. HIV and hepatitis.
* Adolescents / young adults who are unable or unwilling to give informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Men with cholestatic liver conditions including but not restricted to Primary Sclerosing Cholangitis and Primary Biliary Cholangitis.
  Fathers with cholestatic liver conditions including but not restricted to Primary Sclerosing Cholangitis and Primary Biliary Cholangitis and their children aged 16 - 25 yeas of age.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Impact of male cholestasis on DNA methylation patterns in sperm | 01/04/2018
Impact of male cholestasis on small RNA content in sperm | 01/04/2018
Impact of male cholestasis on sperm histone retention | 01/04/2018
Impact of paternal cholestasis on the BMI, hip and waist girth of their adolescent / young adult children | 01/04/2018
Impact of paternal cholestasis on the general health of their adolescent / young adult children | 01/04/2018
  The prevalence of heart, lung, diabetes, thyroid, kidney or liver disease in children of fathers with cholestasis will be investigated

SECONDARY OUTCOMES:
Impact of male cholestasis on seminal fluid composition. | 01/04/2018

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Assisted Conception Unit, Guy's Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No